CLINICAL TRIAL: NCT03876405
Title: Evaluation of a Non-invasive Sensory Feedback System in Hand Prostheses in Everyday Life.
Brief Title: Evaluation of a Non-invasive Sensory Feedback System in Hand Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Ulrika Wijk, Principal Investigator, Lund University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SFB2014
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Amputation, Traumatic; Prosthesis User
Keywords: hand prosthesis; sensory feedback; amputation; upper limb
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sensory feedback (Experimental): A non-invasive air-mediated sensory feedback system embedded in the prosthesis socket.
  Group description: Individuals with acquired forearm amputation.
  Interventions: Device: smartskin non-invasive sensory feedback

INTERVENTIONS:
Device: smartskin non-invasive sensory feedback — The sensory feedback system used was a simple non-invasive, non-electronic system based on air-mediated pressure. A silicone glove with bulbs (35 mm in length) volar in every fingertip was made and applied on a VariPlus Speed hand (OttoBock), size 7¾.
  The sensory feedback system was embedded in the prosthetic socket.

SUMMARY:
Implication and evaluation of a non-invasive sensory feedback system in hand prostheses in everyday life.

DETAILED DESCRIPTION:
A non invasive sensory feedback system in embedded in the prosthetic socket will be tested on forearm amputees in their everday life. Pretests and follow up will contain objective outcome assessments and semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* acquired forearm amputation

Exclusion Criteria:

* psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Assessment of Myoelectric Control - ACMC | 2 days
  An observational assessment where you rate the subjects' capacity of myoelectric control in a bimanual activity. The scoring was made by an experienced external rater.
Task performance questionnaire | 2 days
  21 questions about sensory feedback from the prosthesis, agency, body ownership, performance in activity and phantom limb pain. Self-administered estimation on a 7 grade Likert-scale.
Pointing task | 2 days
  A objective measurement of body ownership. The subject are asked to mark on a ruler, with the hand prosthesis hidden, where they estimate the location of the prosthetic index finger.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wijk U, Carlsson IK, Antfolk C, Bjorkman A, Rosen B. Sensory Feedback in Hand Prostheses: A Prospective Study of Everyday Use. Front Neurosci. 2020 Jul 7;14:663. doi: 10.3389/fnins.2020.00663. eCollection 2020. PMID 32733187